CLINICAL TRIAL: NCT05473819
Title: Effectiveness of Sodium Bicarbonate Buffered Anaesthetic Solution on Pain During Inferior Alveolar Nerve Block in Children : a Randomised Controlled Clinical Trial
Brief Title: Effectiveness of Sodium Bicarbonate Buffered Anaesthetic Solution on Pain During Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2890
Record Dates: First submitted 2022-07-01; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-01

CONDITIONS: Local Anesthesia
Keywords: buffered; sodium bicarbonate; inferior alveolar nerve block; pain; pulpotomy; articaine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Split Mouth Design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buffered Anaesthetic solution (Experimental): 8.4% sodium bicarbonate will be added to the 4% articaine HCL with 1:1000000 epinephrine carpule in ratio 19:1 the Articaine to the Sodium bicarbonate
  Interventions: Drug: Buffered Local Anesthesia
- Conventional Anaesthetic solution (Active Comparator): 4% Articaine HCL with 1:1000000 epinephrine Anaesthetic carpule
  Interventions: Drug: Conventional Unbuffered Local Anesthesia

INTERVENTIONS:
Drug: Buffered Local Anesthesia — Buffered local anesthesia will be administered after being previously prepared just before the injection time.
  Buffering Local Anesthetic Solutions Using 8.4% Sodium Bicarbonate in a 19:1 Ratio: Using the "REMOVE AND REPLACE hand buffering method"
  -Under sterile conditions, 0.09 mL of local anesthetic solution will be removed from the cartridge using a 0.5 mL syringe with a 28- gauge, 0.5-inch needle (Kendall Monoject Insulin Syringe [Tyco Healthcare, tyco.com] lot number 027501). Using a separate unused syringe, 0.09 mL of the commercially available 8.4% sodium bicarbonate will be removed from the 50 mL vial and immediately injected into the local anesthetic cartridge. The cartridge will be inverted 5 times to mix the solution, and no precipitation will be present.
  Arms: Buffered Anaesthetic solution
Drug: Conventional Unbuffered Local Anesthesia — The control group will receive the unbuffered conventional anaesthetic solution
  Arms: Conventional Anaesthetic solution

SUMMARY:
This study will test the effectiveness of addition of Sodium Bicarbonate as a buffering agent to the anaesthetic solution on minimizing the pain of injection and increasing the onset time and potency of the anaesthetic solution in children

DETAILED DESCRIPTION:
27 healthy cooperative children will be enrolled in the study after taking their guardians' informed consent.

The study design will be a split mouth design where each patient will be received buffered anaesthetic solution (8.4% sodium bicarbonate will be added to the anaesthetic solution in ratio 1:19) in one side and conventional anaesthetic solution (4% articaine HCL with 1:1000000 epinephrine) in the other side.

The pain during injection for each patient in both sides will be then compared using objective and subjective methods.

The onset time of the anaesthesia in both sides will also be compared for each patient using Transcutaneous electric nerve stimulator device (TENS)

The results will be collected and mentioned.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 5 - 7 years.
* Children free of any systemic disease or special health care need (ASA I).
* No previous bad dental experience.
* Positive or definitely positive behaviour during preoperative assessments according to the Frankl Rating Scale (score 3 or 4)
* Patients whom their lower primary molars bilaterally are indicated for pulpotomy.
* Patients whom their parents will give consent to participate.
* Patients who give multiple reliable responses while using the transcutaneous electric nerve stimulator device.

Exclusion Criteria:

* Active sites of pathosis in area of injection that could affect anaesthetic assessment.
* History of allergy to local anaesthesia.
* Root resorption affecting more than one third of the root length.
* Fractured crowns due to trauma.
* Clinical signs and symptoms of pulp degeneration such as swelling or sinus tracts
* Radiographic evidence of periapical or interradicular radiolucency
* Non restorable crowns.
* Signs of mobility.
* Ankylosed roots.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain during inferior alveolar nerve block injection | during local anesthesia administration
  Sound, Eye, Motor (SEM) Scale (Appendix II), will be used as an objective method for pain assessment. It comprises the following parameters: (1) Sound, (2) Eye, (3) Motor. For each child, the sounds, eye symptoms and body movements will be evaluated by the operator using the recorded video tapes. The slightest manifestations of the sound, eyes, or motion of the patient is graded in four levels: comfort, mild, moderate, and severe discomfort, and subsequently given grades 1 (comfort), 2 (mild discomfort), 3 (moderate discomfort), and 4 (severe discomfort), respectively. SEM score will be calculated by summing the three grades of the parameters

SECONDARY OUTCOMES:
the onset time of the Anaesthesia | after local anesthesia administration
  Current Perception Threshold (CPT) detection using Transcutaneous Electric Nerve Stimulator (TENS) device. CPT baseline value is the lowest intensity at which the patient first report feeling the stimulus. It determines the Sensory Threshold (ST), which corresponds to the lowest current intensity capable of eliciting perception. The electrode will be placed on the proposed measuring site and the device will be turned on. The device will start the delivery of current at the lowest output intensity and then slowly increased until the patient reported feeling the stimulus. Patients will be instructed to state if they feel any sensation, at that time the delivery of electrical current will be terminated and CPT intensity will be recorded. Every 30 seconds after administration of anaesthesia, while set at the baseline CPT intensity recording for each patient, the electrode will be applied to the proposed measuring site on the anesthetized side, to detect the time of onset of anaesthesia.

OTHER OUTCOMES:
the effectiveness of the anaesthesia | after local anesthesia administration
  This will be determined through completion of the procedure without pain with no need for additional anaesthetic injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Kholoud Mamdouh Ahmed Nour, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the results and the outcomes